CLINICAL TRIAL: NCT02547974
Title: An Observer-blind Study to Evaluate the Safety, Reactogenicity and Immunogenicity of the Investigational GSK Biologicals' GSK3277511A Vaccine in Adults.
Brief Title: A Study to Evaluate the Safety, Reactogenicity and Immunogenicity of the Investigational GSK Biologicals' GSK3277511A Vaccine in Adults.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 201281; 2015-000378-36 (EudraCT Number)
Record Dates: First submitted 2015-08-27; First posted 2015-09-14 (Estimated); Results first posted 2018-07-23 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-03

CONDITIONS: Respiratory Disorders
Keywords: Safety; Immunogenicity; Reactogenicity
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (4):
- GSK3277513A F1 Group (Experimental): Subjects, 18 - 40 years, receiving two doses of the non adjuvanted GSK Biologicals' NTHi Mcat investigational vaccine (GSK3277513A ) containing formulation 1 (F1) of PD, PE-PilA and UspA2 during Step 1 of the study. Intramuscular injection should be done in the deltoid of the non-dominant arm. In case it is not possible to inject in the non dominant arm, an injection in the dominant arm may be performed.
  Interventions: Biological: Formulation 1 (plain): NTHi/Mcat vaccine GSK3277513A
- GSK3277513A F2 Group (Experimental): Subjects, 50 - 70 years, receiving two doses of the GSK Biologicals' NTHi-Mcat investigational vaccine(GSK3277513A) containing formulation 2 (F2) (adjuvanted) of PD, PE-PilA and UspA2 during Step 2 of the study. Intramuscular injection should be done in the deltoid of the non-dominant arm. In case it is not possible to inject in the non dominant arm, an injection in the dominant arm may be performed.
  Interventions: Biological: Formulation 2 (adjuvanted): NTHi/Mcat vaccine GSK3277513A
- GSK3277513A F3 Group (Experimental): Subjects, 50 - 70 years, receiving two doses of the GSK Biologicals' NTHi-Mcat investigational vaccine(GSK3277513A) containing formulation 3 (F3) (adjuvanted) of PD, PE-PilA and UspA2 during Step 2 of the study. Intramuscular injection should be done in the deltoid of the non-dominant arm. In case it is not possible to inject in the non dominant arm, an injection in the dominant arm may be performed.
  Interventions: Biological: Formulation 3 (adjuvanted): NTHi/Mcat vaccine GSK3339036A
- Placebo Group (Placebo Comparator): Subjects, 18 - 40 years, receiving two doses of placebo (saline solution) during Step 1 of the study and subjects, 50 - 70 years, receiving two doses of placebo (saline solution) during Step 2 of the study. Intramuscular injection should be done in the deltoid of the non-dominant arm. In case it is not possible to inject in the non dominant arm, an injection in the dominant arm may be performed.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Formulation 1 (plain): NTHi/Mcat vaccine GSK3277513A — 2 doses at Day 0 and Day 60, Intramuscular vaccination in the deltoid region of the non-dominant arm according to protocol schedule
  Arms: GSK3277513A F1 Group
Biological: Formulation 2 (adjuvanted): NTHi/Mcat vaccine GSK3277513A — 2 doses at Day 0 and Day 60, Intramuscular vaccination in the deltoid region of the non-dominant arm according to protocol schedule
  Arms: GSK3277513A F2 Group
Biological: Formulation 3 (adjuvanted): NTHi/Mcat vaccine GSK3339036A — 2 doses at Day 0 and Day 60, Intramuscular vaccination in the deltoid region of the non-dominant arm according to protocol schedule
  Arms: GSK3277513A F3 Group
Drug: Placebo — 2 doses at Day 0 and Day 60, Intramuscular vaccination in the deltoid region of the non-dominant arm according to protocol schedule
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to assess the safety, reactogenicity and immunogenicity of the investigational GSK Biologicals' GSK3277511A vaccine in adults

ELIGIBILITY:
Inclusion Criteria:

applicable for both Step 1 ((healthy volunteers) and Step 2 ([ex-]smokers)

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol
* Written informed consent obtained from the subject.
* Female subjects of non-childbearing potential may be enrolled in the study.

  * Non-childbearing potential is defined as pre-menarche, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vacci-nation, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

only applicable for Step 1

* A male or female between, and including, 18 and 40 years of age at the time of the Screening Visit.
* Healthy subjects without acute or chronic, clinically sig-nificant pulmonary, cardiovascular, hepatic or renal func-tional abnormality, as determined by physical examination or laboratory screening tests.

only applicable for Step 2

* A male or female between, and including, 50 and 70 years of age at the time of the screening visit.
* Subjects without medical history, clinical finding or laboratory finding which in the opinion of the investigator could pose a safety concern or interfere with the protocol.
* Current or former smoker with a cigarette smoking history ≥ 10 pack-years.

Exclusion Criteria:

applicable for both Step 1 and Step 2

* Use of any investigational or non-registered product other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product.
* Previous vaccination with any vaccine containing NTHi and/or Mcat antigens.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs within 6 months prior to the first vaccine dose. For corticosteroids, this will mean prednisone ≥20 mg/day, or equivalent. Only topical steroids are allowed.
* Administration of long-acting immune-modifying drugs at any time during the study period.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the first dose of study vaccine or planned administration during the study period.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of or current autoimmune disease.
* Acute disease and/or fever at the time of enrolment.

  * Fever is defined as temperature >= 37.5°C for oral or axillary route. The preferred route for recording temperature in this study will be oral.
  * Subjects with a minor illness without fever may, be enrolled at the discretion of the investigator.
* Current alcoholism and/or drug abuse.
* History of or current condition preventing intramuscular injection as bleeding or coagulation disorder.
* Malignancies within previous 5 years or lymphoproliferative disorders.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* Any other condition that the investigator judges may interfere with study findings.

only applicable for Step 1

* Planned administration/ administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the first dose and ending 30 days after the last dose of vaccine, with the exception of any influenza vaccine which may be administered ≥ 15 days preceding or following any study vaccine dose.
* Laboratory evidence of clinically significant haematological (complete blood cell count [RBC, WBC], WBC differential count [lymphocytes, neutrophils and eosinophils], platelets count or haemoglobin level) and biochemical (alanine aminotransferase [ALT], aspartate aminotransferase [AST] or creatinine) abnormalities as per the opinion of the investigator.

only applicable for Step 2

* Planned administration/ administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the first dose and ending 30 days after the last dose of vaccine, with the exception of any influenza or pneumococcal licensed vaccine which may be admin-istered ≥ 15 days preceding or following any study vaccine dose.
* Post-bronchodilator FEV1 < 80% of predicted normal value.
* Diagnosed with a respiratory disorder (e.g. asthma, COPD, sarcoidosis, tuberculosis, bronchiectasis, lung fi-brosis, pulmonary embolism, pneumothorax, or physi-cian confirmed lung cancer). Please note that subjects with mild pulmonary obstruction (i.e. FEV1/ FVC ratio < 0.7 with FEV1 ≥ 80% of normal predicted values [GOLD grade 1]) can be enrolled.
* Has contraindication for spirometry testing (such as recent eye surgery, recent thoracic or abdominal surgery procedures, unstable cardiovascular status, recent myo-cardial infection or pulmonary embolism).
* Laboratory evidence of clinically significant haematological (complete blood cell count [RBC, WBC], WBC differential count [lymphocytes, neutrophils and eosinophils], platelets count or haemoglobin level) and biochemical (ALT, AST or creatinine) abnormalities.
* Has significant disease, in the opinion of the investigator, likely to interfere with the study and/or likely to cause death within the study duration.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-08-31 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Belgium (3):
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Wilrijk

REFERENCES:
- [Derived] Van Damme P, Leroux-Roels G, Vandermeulen C, De Ryck I, Tasciotti A, Dozot M, Moraschini L, Testa M, Arora AK. Safety and immunogenicity of non-typeable Haemophilus influenzae-Moraxella catarrhalis vaccine. Vaccine. 2019 May 21;37(23):3113-3122. doi: 10.1016/j.vaccine.2019.04.041. Epub 2019 Apr 24. PMID 31029515

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 120 subjects were enrolled in the study. All subjects received at least one dose of the vaccine.
Pre-assignment Details: For each subject, the study lasted approximately 15 months, from screening (Pre-Day 0) to study end (Day 420). Vaccination schedules: 0, 2 months (i.e. at Day 0 and Day 60).
Period: Overall Study
Arm/Group | GSK3277513A F1 Group | GSK3277513A F2 Group | GSK3277513A F3 Group | PLACEBO Group
Started | 15 | 31 | 30 | 44
Completed | 14 | 31 | 30 | 44
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK3277513A F1 Group | GSK3277513A F2 Group | GSK3277513A F3 Group | PLACEBO Group | Total
Number analyzed (Participants) | 15 | 31 | 30 | 44 | 120
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.1 (5.91) | 58.9 (6.49) | 58.5 (5.82) | 47.2 (16.72) | 50.8 (14.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 13 | 21 | 58
  Male | 4 | 18 | 17 | 23 | 62
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - Caucasian / European Heritage | 15 | 31 | 30 | 44 | 120

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Any Solicited Local Adverse Events (AEs)
Description: Assessed solicited local symptoms are pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: During a 7-day follow-up period (Day 0 to Day 6) after first dose.
Population: Analysis was performed on the total vaccinated cohort which included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3277513A F1 Group | GSK3277513A F2 Group | GSK3277513A F3 Group | PLACEBO Group
Number analyzed (Participants) | 15 | 31 | 30 | 44
Participants
  Any Pain | 2 | 19 | 26 | 6
  Any Redness (mm) | 0 | 3 | 2 | 0
  Any Swelling (mm) | 0 | 4 | 0 | 0

2. Primary Outcome: Number of Subjects With Any Solicited Local Adverse Events (AEs)
Description: as for outcome 1
Time Frame: During a 7-day follow-up period (Day 60 to Day 66) after second dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3277513A F1 Group | GSK3277513A F2 Group | GSK3277513A F3 Group | PLACEBO Group
Number analyzed (Participants) | 14 | 31 | 29 | 44
Participants
  Any Pain | 7 | 23 | 25 | 8
  Any Redness (mm) | 0 | 3 | 4 | 0
  Any Swelling (mm) | 0 | 2 | 3 | 0

3. Primary Outcome: Number of Subjects With Any Solicited General Adverse Events (AEs)
Description: Assessed solicited general symptoms are fatigue, gastrointestinal symptoms, headache, myalgia, fever [defined as oral temperature equal to or above 37.5 degrees Celsius (°C)].
Time Frame: During a 7-day follow-up period (Day 0 to Day 6) after first dose.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3277513A F1 Group | GSK3277513A F2 Group | GSK3277513A F3 Group | PLACEBO Group
Number analyzed (Participants) | 15 | 31 | 30 | 44
Participants
  Any Fatigue | 3 | 3 | 11 | 10
  Any Gastrointestinal symptoms | 1 | 0 | 4 | 3
  Any Headache | 4 | 2 | 10 | 7
  Any Myalgia | 2 | 6 | 7 | 4
  Any Temperature (Oral) (°C) | 1 | 0 | 2 | 0

4. Primary Outcome: Number of Subjects With Any Solicited General Adverse Events (AEs)
Description: as for outcome 3
Time Frame: During a 7-day follow-up period (Day 60 to Day 66) after second dose.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3277513A F1 Group | GSK3277513A F2 Group | GSK3277513A F3 Group | PLACEBO Group
Number analyzed (Participants) | 14 | 31 | 29 | 44
Participants
  Any Fatigue | 3 | 9 | 13 | 6
  Any Gastrointestinal symptoms | 3 | 2 | 3 | 1
  Any Headache | 3 | 5 | 8 | 2
  Any Myalgia | 1 | 9 | 8 | 3
  Any Temperature (Oral) (°C) | 0 | 3 | 3 | 1

5. Primary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs).
Description: Assessed unsolicited AEs cover any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any is defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During a 30-day follow-up period (Day 0 to Day 29) after first dose.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3277513A F1 Group | GSK3277513A F2 Group | GSK3277513A F3 Group | PLACEBO Group
Number analyzed (Participants) | 15 | 31 | 30 | 44
Participants | 6 | 13 | 14 | 21

6. Primary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: as for outcome 5
Time Frame: During a 30-day follow-up period (Day 60 to Day 89) after second dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3277513A F1 Group | GSK3277513A F2 Group | GSK3277513A F3 Group | PLACEBO Group
Number analyzed (Participants) | 15 | 31 | 30 | 44
Participants | 6 | 14 | 14 | 19

7. Primary Outcome: Number of Subjects With Any Haematological and Biochemical Laboratory Abnormalities, After Vaccination.
Description: Assessed haematological parameters are complete blood cell count: Erythrocytes (RBC [red blood cells]), Leukocytes (WBC [white blood cells]), differential count (basophils, eosinophils, lymphocytes, monocytes, neutrophils), platelets count, and hemoglobin level below or above the normal laboratory ranges tabulated by time point.
  Assessed biochemical parameters are alanine aminotransferase [ALT], aspartate aminotransferase [AST] or creatinine below or above the normal laboratory ranges tabulated by time point.
Time Frame: At Day 7, post-dose 1.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3277513A F1 Group | GSK3277513A F2 Group | GSK3277513A F3 Group | PLACEBO Group
Number analyzed (Participants) | 15 | 31 | 30 | 44
Participants
  ALT below: number analyzed (Participants) | 15 | 30 | 30 | 44
  ALT below | 0 | 0 | 0 | 0
  ALT above: number analyzed (Participants) | 15 | 30 | 30 | 44
  ALT above | 0 | 0 | 0 | 3
  AST below: number analyzed (Participants) | 15 | 30 | 30 | 44
  AST below | 0 | 0 | 0 | 0
  AST above: number analyzed (Participants) | 15 | 30 | 30 | 44
  AST above | 0 | 0 | 0 | 1
  Basophils below | 0 | 0 | 0 | 0
  Basophils above | 0 | 0 | 0 | 0
  Creatinine below: number analyzed (Participants) | 15 | 30 | 30 | 44
  Creatinine below | 0 | 1 | 2 | 1
  Creatinine above: number analyzed (Participants) | 15 | 30 | 30 | 44
  Creatinine above | 1 | 1 | 0 | 1
  Eosinophils below | 2 | 2 | 0 | 0
  Eosinophils above | 0 | 0 | 1 | 1
  Erythrocytes below | 0 | 0 | 2 | 3
  Erythrocytes above | 0 | 2 | 1 | 1
  Hemoglobin below | 0 | 1 | 4 | 4
  Hemoglobin above | 0 | 0 | 0 | 0
  Leucocytes below | 0 | 1 | 0 | 0
  Leucocytes above | 0 | 3 | 1 | 1
  Lymphocytes below | 0 | 0 | 0 | 0
  Lymphocytes above | 0 | 0 | 0 | 0
  Monocytes below | 2 | 1 | 0 | 1
  Monocytes above | 1 | 0 | 0 | 0
  Neutrophils below | 1 | 0 | 0 | 0
  Neutrophils above | 0 | 3 | 0 | 1
  Platelets below | 0 | 0 | 0 | 0
  Platelets above | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Subjects With Any Haematological and Biochemical Laboratory Abnormalities After Vaccination
Description: as for outcome 7
Time Frame: At Day 60, post-dose 1.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3277513A F1 Group | GSK3277513A F2 Group | GSK3277513A F3 Group | PLACEBO Group
Number analyzed (Participants) | 14 | 31 | 30 | 44
Participants
  ALT below | 0 | 0 | 0 | 0
  ALT above | 0 | 1 | 0 | 1
  AST below | 0 | 0 | 0 | 0
  AST above | 0 | 1 | 0 | 1
  Basophils below: number analyzed (Participants) | 14 | 29 | 28 | 41
  Basophils below | 0 | 0 | 0 | 0
  Basophils above: number analyzed (Participants) | 14 | 29 | 28 | 41
  Basophils above | 0 | 0 | 0 | 0
  Creatinine below | 0 | 1 | 3 | 2
  Creatinine above | 1 | 1 | 0 | 1
  Eosinophils below: number analyzed (Participants) | 14 | 29 | 28 | 41
  Eosinophils below | 5 | 2 | 1 | 2
  Eosinophils above: number analyzed (Participants) | 14 | 29 | 28 | 41
  Eosinophils above | 1 | 0 | 1 | 0
  Erythrocytes below: number analyzed (Participants) | 14 | 29 | 28 | 41
  Erythrocytes below | 0 | 0 | 1 | 1
  Erythrocytes above: number analyzed (Participants) | 14 | 29 | 28 | 41
  Erythrocytes above | 0 | 1 | 1 | 1
  Hemoglobin below: number analyzed (Participants) | 14 | 29 | 28 | 41
  Hemoglobin below | 1 | 0 | 2 | 3
  Hemoglobin above: number analyzed (Participants) | 14 | 29 | 28 | 41
  Hemoglobin above | 0 | 1 | 1 | 0
  Leucocytes below: number analyzed (Participants) | 14 | 29 | 28 | 41
  Leucocytes below | 0 | 0 | 1 | 0
  Leucocytes above: number analyzed (Participants) | 14 | 29 | 28 | 41
  Leucocytes above | 0 | 1 | 0 | 1
  Lymphocytes below: number analyzed (Participants) | 14 | 29 | 28 | 41
  Lymphocytes below | 0 | 1 | 0 | 0
  Lymphocytes above: number analyzed (Participants) | 14 | 29 | 28 | 41
  Lymphocytes above | 0 | 0 | 0 | 0
  Monocytes below: number analyzed (Participants) | 14 | 29 | 28 | 41
  Monocytes below | 0 | 0 | 1 | 0
  Monocytes above: number analyzed (Participants) | 14 | 29 | 28 | 41
  Monocytes above | 0 | 0 | 0 | 0
  Neutrophils below: number analyzed (Participants) | 14 | 29 | 28 | 41
  Neutrophils below | 0 | 0 | 0 | 0
  Neutrophils above: number analyzed (Participants) | 14 | 29 | 28 | 41
  Neutrophils above | 0 | 1 | 0 | 0
  Platelets below: number analyzed (Participants) | 14 | 29 | 28 | 41
  Platelets below | 0 | 0 | 1 | 0
  Platelets above: number analyzed (Participants) | 14 | 29 | 28 | 41
  Platelets above | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Subjects With Any Haematological and Biochemical Laboratory Abnormalities After Vaccination
Description: as for outcome 7
Time Frame: At Day 67, post-dose 2.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3277513A F1 Group | GSK3277513A F2 Group | GSK3277513A F3 Group | PLACEBO Group
Number analyzed (Participants) | 14 | 31 | 30 | 44
Participants
  ALT below | 0 | 0 | 0 | 0
  ALT above | 0 | 1 | 1 | 1
  AST below | 0 | 0 | 0 | 0
  AST above | 0 | 0 | 0 | 2
  Basophils below | 0 | 0 | 0 | 0
  Basophils above | 0 | 0 | 0 | 0
  Creatinine below | 1 | 1 | 1 | 1
  Creatinine above | 1 | 2 | 0 | 1
  Eosinophils below | 1 | 0 | 1 | 2
  Eosinophils above | 0 | 0 | 1 | 1
  Erythrocytes below | 0 | 1 | 1 | 2
  Erythrocytes above | 0 | 1 | 1 | 1
  Hemoglobin below | 1 | 3 | 1 | 3
  Hemoglobin above | 0 | 0 | 0 | 0
  Leucocytes below | 0 | 0 | 0 | 0
  Leucocytes above | 0 | 4 | 1 | 1
  Lymphocytes below | 0 | 0 | 1 | 0
  Lymphocytes above | 0 | 1 | 0 | 0
  Monocytes below | 0 | 0 | 0 | 0
  Monocytes above | 0 | 0 | 1 | 0
  Neutrophils below | 0 | 1 | 0 | 0
  Neutrophils above | 0 | 3 | 1 | 1
  Platelets below | 0 | 0 | 1 | 0
  Platelets above | 0 | 0 | 0 | 0

10. Primary Outcome: Number of Subjects With Any Haematological and Biochemical Laboratory Abnormalities After Vaccination
Description: as for outcome 7
Time Frame: At Day 210, post-dose 2.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3277513A F1 Group | GSK3277513A F2 Group | GSK3277513A F3 Group | PLACEBO Group
Number analyzed (Participants) | 14 | 31 | 30 | 44
Participants
  ALT below | 0 | 0 | 0 | 0
  ALT above | 0 | 2 | 1 | 1
  AST below | 0 | 0 | 0 | 0
  AST above | 0 | 1 | 1 | 0
  Basophils below: number analyzed (Participants) | 14 | 31 | 30 | 43
  Basophils below | 0 | 0 | 0 | 0
  Basophils above: number analyzed (Participants) | 14 | 31 | 30 | 43
  Basophils above | 0 | 0 | 0 | 0
  Creatinine below | 0 | 2 | 2 | 2
  Creatinine above | 1 | 1 | 0 | 1
  Eosinophils below: number analyzed (Participants) | 14 | 31 | 30 | 43
  Eosinophils below | 4 | 2 | 3 | 4
  Eosinophils above: number analyzed (Participants) | 14 | 31 | 30 | 43
  Eosinophils above | 0 | 0 | 1 | 0
  Erythrocytes below | 1 | 1 | 1 | 1
  Erythrocytes above | 0 | 1 | 1 | 0
  Hemoglobin below | 2 | 2 | 1 | 6
  Hemoglobin above | 0 | 0 | 0 | 0
  Leucocytes below | 0 | 0 | 0 | 0
  Leucocytes above | 0 | 2 | 0 | 1
  Lymphocytes below: number analyzed (Participants) | 14 | 31 | 30 | 43
  Lymphocytes below | 0 | 2 | 0 | 0
  Lymphocytes above: number analyzed (Participants) | 14 | 31 | 30 | 43
  Lymphocytes above | 0 | 0 | 0 | 1
  Monocytes below: number analyzed (Participants) | 14 | 31 | 30 | 43
  Monocytes below | 1 | 2 | 1 | 2
  Monocytes above: number analyzed (Participants) | 14 | 31 | 30 | 43
  Monocytes above | 0 | 0 | 0 | 0
  Neutrophils below: number analyzed (Participants) | 14 | 31 | 30 | 43
  Neutrophils below | 0 | 0 | 0 | 0
  Neutrophils above: number analyzed (Participants) | 14 | 31 | 30 | 43
  Neutrophils above | 0 | 2 | 1 | 1
  Platelets below | 0 | 0 | 1 | 0
  Platelets above | 0 | 0 | 0 | 0

11. Primary Outcome: Number of Subjects With Any Haematological and Biochemical Laboratory Abnormalities After Vaccination
Description: as for outcome 7
Time Frame: At Day 420, post-dose 2.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3277513A F1 Group | GSK3277513A F2 Group | GSK3277513A F3 Group | PLACEBO Group
Number analyzed (Participants) | 14 | 31 | 30 | 44
Participants
  ALT below | 0 | 0 | 0 | 0
  ALT above | 0 | 1 | 0 | 1
  AST below | 0 | 0 | 0 | 0
  AST above | 0 | 1 | 0 | 0
  Basophils below: number analyzed (Participants) | 14 | 31 | 29 | 44
  Basophils below | 0 | 0 | 0 | 0
  Basophils above: number analyzed (Participants) | 14 | 31 | 29 | 44
  Basophils above | 0 | 0 | 0 | 0
  Creatinine below | 1 | 1 | 2 | 3
  Creatinine above | 0 | 1 | 0 | 0
  Eosinophils below: number analyzed (Participants) | 14 | 31 | 29 | 44
  Eosinophils below | 4 | 0 | 1 | 2
  Eosinophils above: number analyzed (Participants) | 14 | 31 | 29 | 44
  Eosinophils above | 0 | 1 | 0 | 1
  Erythrocytes below: number analyzed (Participants) | 14 | 31 | 29 | 44
  Erythrocytes below | 0 | 0 | 1 | 2
  Erythrocytes above: number analyzed (Participants) | 14 | 31 | 29 | 44
  Erythrocytes above | 0 | 1 | 1 | 0
  Hemoglobin below: number analyzed (Participants) | 14 | 31 | 29 | 44
  Hemoglobin below | 0 | 1 | 0 | 2
  Hemoglobin above: number analyzed (Participants) | 14 | 31 | 29 | 44
  Hemoglobin above | 0 | 1 | 0 | 1
  Leucocytes below: number analyzed (Participants) | 14 | 31 | 29 | 44
  Leucocytes below | 0 | 0 | 0 | 0
  Leucocytes above: number analyzed (Participants) | 14 | 31 | 29 | 44
  Leucocytes above | 0 | 3 | 1 | 1
  Lymphocytes below: number analyzed (Participants) | 14 | 31 | 29 | 44
  Lymphocytes below | 0 | 1 | 0 | 0
  Lymphocytes above: number analyzed (Participants) | 14 | 31 | 29 | 44
  Lymphocytes above | 0 | 0 | 0 | 0
  Monocytes below: number analyzed (Participants) | 14 | 31 | 29 | 44
  Monocytes below | 3 | 0 | 0 | 1
  Monocytes above: number analyzed (Participants) | 14 | 31 | 29 | 44
  Monocytes above | 0 | 0 | 0 | 1
  Neutrophils below: number analyzed (Participants) | 14 | 31 | 29 | 44
  Neutrophils below | 0 | 1 | 1 | 1
  Neutrophils above: number analyzed (Participants) | 14 | 31 | 29 | 44
  Neutrophils above | 0 | 3 | 1 | 1
  Platelets below: number analyzed (Participants) | 14 | 31 | 29 | 44
  Platelets below | 0 | 0 | 1 | 0
  Platelets above: number analyzed (Participants) | 14 | 31 | 29 | 44
  Platelets above | 0 | 0 | 0 | 0

12. Primary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs)
Description: Assessed SAEs include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From first vaccination up to study conclusion (Day 0 to Day 420)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3277513A F1 Group | GSK3277513A F2 Group | GSK3277513A F3 Group | PLACEBO Group
Number analyzed (Participants) | 15 | 31 | 30 | 44
Participants | 1 | 0 | 1 | 2

13. Primary Outcome: Number of Subjects With Any Potential Immune-mediated Diseases (pIMDs)
Description: Potential immune-mediated diseases (pIMDs) are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
Time Frame: From first vaccination up to study conclusion (Day 0 to Day 420)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3277513A F1 Group | GSK3277513A F2 Group | GSK3277513A F3 Group | PLACEBO Group
Number analyzed (Participants) | 15 | 31 | 30 | 44
Participants | 1 | 0 | 1 | 0

14. Secondary Outcome: Concentration of Antibodies Against the NTHi-Mcat Anti-PD (Protein D of Haemophilus Influenzae) Vaccine Component
Description: Antibody concentrations are measured by enzyme-linked immunosorbent assay (ELISA) and expressed as geometric mean concentrations (GMCs) in ELISA units per millilitre (EL.U/mL). The cut-off of the assay is 153 EL.U/mL for anti-PD antibodies.
Time Frame: At Day 0 (pre-dose 1); at Day 30 and Day 60 (post-dose 1); at Day 90, Day 210 and Day 420 (post-dose2).
Population: The analysis was performed on the According-to-Protocol cohort for immunogenicity, which included all evaluable subjects (i.e. those meeting all eligibility criteria, complying with the procedures defined in the protocol, with no elimination criteria during the study) for whom data concerning immunogenicity outcome variables were available.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | GSK3277513A F1 Group | GSK3277513A F2 Group | GSK3277513A F3 Group | PLACEBO Group
Number analyzed (Participants) | 14 | 31 | 29 | 43
EL.U/mL
  Anti-PD antibody, Day 0: number analyzed (Participants) | 14 | 30 | 29 | 43
  Anti-PD antibody, Day 0 | 109.7 [71.2 to 169.1] | 102.8 [77.5 to 136.4] | 88.1 [72.4 to 107.1] | 89 [75 to 105.7]
  Anti-PD antibody, Day 30 | 239.8 [123 to 467.6] | 569.4 [335.9 to 965.3] | 818 [532 to 1257.8] | 90.8 [76.5 to 107.8]
  Anti-PD antibody, Day 60: number analyzed (Participants) | 14 | 30 | 29 | 43
  Anti-PD antibody, Day 60 | 220.9 [121.1 to 402.9] | 327.1 [207.4 to 515.6] | 495 [307.2 to 797.5] | 88.6 [75.2 to 104.3]
  Anti-PD antibody, Day 90 | 289.2 [144.6 to 578.5] | 984.4 [662.3 to 1463.2] | 1538.5 [1134.6 to 2086.2] | 91.8 [77.8 to 108.3]
  Anti-PD antibody, Day 210 | 179.5 [96.7 to 333.5] | 471.8 [310.2 to 717.5] | 806.1 [560.2 to 1159.9] | 92.9 [79 to 109.2]
  Anti-PD antibody, Day 420 | 165.1 [89.7 to 303.8] | 370.2 [238.2 to 575.3] | 538.1 [369.1 to 784.5] | 88.8 [77.3 to 102.1]

15. Secondary Outcome: Concentration of Antibodies Against the NTHi-Mcat Anti-PE (Protein E of Haemophilus Influenzae) Vaccine Component
Description: Antibody concentrations are measured by enzyme-linked immunosorbent assay (ELISA) and expressed as geometric mean concentrations (GMCs) in ELISA units per millilitre (EL.U/mL). The cut-off of the assay is 25 EL.U/mL for anti-PE antibodies.
Time Frame: At Day 0 (pre-dose 1); at Day 30 and Day 60 (post-dose 1); at Day 90, Day 210 and Day 420 (post-dose2).
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | GSK3277513A F1 Group | GSK3277513A F2 Group | GSK3277513A F3 Group | PLACEBO Group
Number analyzed (Participants) | 14 | 31 | 29 | 43
EL.U/mL
  Anti-PE antibody, Day 0 | 31.3 [16.4 to 59.7] | 20.6 [15.7 to 27] | 19.7 [14.8 to 26.2] | 21.9 [17 to 28.1]
  Anti-PE antibody, Day 30: number analyzed (Participants) | 13 | 31 | 29 | 43
  Anti-PE antibody, Day 30 | 178.3 [64.6 to 491.9] | 627.2 [401 to 980.9] | 1287.8 [816.2 to 2032] | 21.3 [16.7 to 27.1]
  Anti-PE antibody, Day 60 | 151.9 [58 to 397.6] | 573.1 [360.1 to 912.1] | 1207.1 [753.8 to 1932.9] | 20.3 [15.9 to 25.9]
  Anti-PE antibody, Day 90 | 719.1 [357.4 to 1446.8] | 5945.2 [4069.5 to 8685.5] | 8983.9 [7150.4 to 11287.5] | 21.8 [17.1 to 27.8]
  Anti-PE antibody, Day 210 | 385.8 [191.2 to 778.4] | 2390.9 [1655.4 to 3453.1] | 3247.6 [2285.2 to 4615.3] | 20.7 [16.5 to 26]
  Anti-PE antibody, Day 420 | 244.1 [112.4 to 529.9] | 1206.6 [817.5 to 1781] | 1701 [1192.1 to 2427.1] | 22.8 [17.5 to 29.7]

16. Secondary Outcome: Concentration of Antibodies Against the NTHi-Mcat Anti-PilA (Type IV Pili Subunit of Non-typeable Haemophilus Influenzae) Vaccine Component
Description: Antibody concentrations are measured by enzyme-linked immunosorbent assay (ELISA) and expressed as geometric mean concentrations (GMCs) in ELISA units per millilitre (EL.U/mL). The cut-off of the assay is 7 EL.U/mL for anti-PilA antibodies.
Time Frame: At Day 0 (pre-dose 1); at Day 30 and Day 60 (post-dose 1); at Day 90 (post-dose2).
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | GSK3277513A F1 Group | GSK3277513A F2 Group | GSK3277513A F3 Group | PLACEBO Group
Number analyzed (Participants) | 14 | 31 | 29 | 43
EL.U/mL
  Anti-PilA antibody, Day 0 | 11.6 [5.3 to 25.2] | 13.5 [8 to 22.6] | 17.1 [11 to 26.5] | 8.8 [6.1 to 12.6]
  Anti-PilA antibody, Day 30: number analyzed (Participants) | 14 | 29 | 29 | 42
  Anti-PilA antibody, Day 30 | 37.2 [13.6 to 101.5] | 238.6 [123.1 to 462.5] | 330.9 [211.7 to 517.2] | 9.2 [6.4 to 13.3]
  Anti-PilA antibody, Day 60: number analyzed (Participants) | 14 | 30 | 29 | 43
  Anti-PilA antibody, Day 60 | 33.2 [11.3 to 97.9] | 177 [83.4 to 375.7] | 321.2 [210.1 to 491.2] | 9 [6.3 to 13]
  Anti-PilA antibody, Day 90: number analyzed (Participants) | 14 | 31 | 29 | 39
  Anti-PilA antibody, Day 90 | 165.8 [76.7 to 358.4] | 1127.5 [751 to 1692.8] | 1722.3 [1383.4 to 2144.2] | 8.6 [5.8 to 12.6]

17. Secondary Outcome: Concentration of Antibodies Against the NTHi-Mcat Anti-PilA (Type IV Pili Subunit of Non-typeable Haemophilus Influenzae) Vaccine Component
Description: Antibody concentrations are measured by enzyme-linked immunosorbent assay (ELISA) and expressed as geometric mean concentrations (GMCs) in ELISA units per millilitre (EL.U/mL). The cut-off of the assay is 16 EL.U/mL for anti-PilA antibodies.
Time Frame: At Day 210 and Day 420 (post-dose2).
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | GSK3277513A F1 Group | GSK3277513A F2 Group | GSK3277513A F3 Group | PLACEBO Group
Number analyzed (Participants) | 14 | 31 | 29 | 43
EL.U/mL
  Anti-PilA antibody, Day 210 | 52 [18.4 to 146.8] | 367.2 [220.2 to 612.3] | 671 [508.6 to 885.2] | 11.5 [9 to 14.8]
  Anti-PilA antibody, Day 420 | 40.8 [16.5 to 100.7] | 181.8 [108 to 305.9] | 322.2 [233.4 to 444.9] | 11.9 [9.2 to 15.5]

18. Secondary Outcome: Concentration of Antibodies Against the NTHi-Mcat Anti-UspA2 (Ubiquitous Surface Protein A2 of Moraxella Catarrhalis) Vaccine Component
Description: Antibody concentrations are measured by enzyme-linked immunosorbent assay (ELISA) and expressed as geometric mean concentrations (GMCs) in ELISA units per millilitre (EL.U/mL). The cut-off of the assay is 38 EL.U/mL for anti-UspA2 antibodies.
Time Frame: At Day 0 (pre-dose 1); at Day 30 and Day 60 (post-dose 1); at Day 90, Day 210 and Day 420 (post-dose2).
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | GSK3277513A F1 Group | GSK3277513A F2 Group | GSK3277513A F3 Group | PLACEBO Group
Number analyzed (Participants) | 14 | 31 | 29 | 43
EL.U/mL
  Anti-UspA2 IgG antibody, Day 0 | 572.5 [254.4 to 1288.6] | 384.1 [253 to 583.2] | 468.1 [330.6 to 662.8] | 548.3 [399.4 to 752.8]
  Anti-UspA2 IgG antibody, Day 30 | 879.9 [396.6 to 1952.4] | 1006.7 [732.5 to 1383.6] | 913.5 [693.3 to 1203.7] | 571.5 [416.9 to 783.4]
  Anti-UspA2 IgG antibody, Day 60 | 780.7 [365.4 to 1668.3] | 754.4 [533.1 to 1067.6] | 714.7 [538.9 to 947.8] | 567 [418 to 769.1]
  Anti-UspA2 IgG antibody, Day 90 | 1172 [654.7 to 2097.9] | 1440.7 [1065.8 to 1947.5] | 1279 [1026.1 to 1594.4] | 621.5 [449.1 to 860]
  Anti-UspA2 IgG antibody, Day 210 | 775.1 [361.3 to 1662.8] | 882.5 [629.8 to 1236.7] | 767.2 [584.8 to 1006.5] | 525.7 [386.8 to 714.5]
  Anti-UspA2 IgG antibody, Day 420 | 732 [339.2 to 1579.5] | 703.6 [501.8 to 986.5] | 673.4 [504.3 to 899.2] | 552.9 [399.7 to 764.9]

19. Secondary Outcome: Frequency of Specific Cluster of Differentiation (CD)4+ T-cells Against NTHi-Mcat Antigens Collected for the Evaluation of Cell-mediated Immune Response
Description: Frequency of specific CD4+ T-cells are measured by flow cytometry intracellular cytokine staining (ICS) expressing two or more markers (such as Interleukin [IL]-2, IL-13, IL-17, Interferon gamma [FN-γ], Tumour necrosis factor alpha [TNF-α] and CD40L). The frequency of specific CD4+ T-cells are summarised [descriptive statistics: Mean and standard deviation (SD)] against each antigen (PD, PE, PilA and UspA2), by group in Step 2 at each time point during which blood samples are collected for CMI.
Time Frame: At Day 0 (pre-dose 1); at Day 60 (post-dose 1); at Day 90, Day 210 and Day 420 (post-dose2).
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: CD4+ T-cells/million cells
Arm/Group | GSK3277513A F2 Group | GSK3277513A F3 Group | PLACEBO Group
Number analyzed (Participants) | 16 | 12 | 15
CD4+ T-cells/million cells
  CD4+.PD, Day 0: number analyzed (Participants) | 12 | 12 | 13
  CD4+.PD, Day 0 | 28.3 (42.1) | 81.8 (92.29) | 37.4 (46.29)
  CD4+.PD, Day 60 | 105.4 (123.95) | 107.8 (117.92) | 55 (91.94)
  CD4+.PD, Day 90: number analyzed (Participants) | 16 | 11 | 13
  CD4+.PD, Day 90 | 283.3 (236.93) | 349.9 (216.5) | 90.5 (117.41)
  CD4+.PD, Day 210: number analyzed (Participants) | 11 | 11 | 13
  CD4+.PD, Day 210 | 120.4 (99.23) | 176.9 (101.39) | 78.7 (112.16)
  CD4+.PD, Day 420: number analyzed (Participants) | 13 | 9 | 14
  CD4+.PD, Day 420 | 154.3 (165.98) | 164.8 (123.33) | 60.3 (82.01)
  CD4+.PE, Day 0: number analyzed (Participants) | 12 | 12 | 13
  CD4+.PE, Day 0 | 89.2 (199.87) | 41.4 (48.55) | 47.1 (70.65)
  CD4+.PE, Day 60 | 370.7 (372.5) | 176.9 (172.74) | 50.9 (47.91)
  CD4+.PE, Day 90: number analyzed (Participants) | 16 | 11 | 13
  CD4+.PE, Day 90 | 1182.2 (1507.29) | 732.7 (804.67) | 52.4 (56.2)
  CD4+.PE, Day 210: number analyzed (Participants) | 12 | 11 | 14
  CD4+.PE, Day 210 | 469.1 (381.87) | 337.4 (228.12) | 39.1 (65.14)
  CD4+.PE, Day 420: number analyzed (Participants) | 14 | 10 | 14
  CD4+.PE, Day 420 | 545 (735.89) | 215.8 (137.79) | 26.6 (51.74)
  CD4+.PilA, Day 0: number analyzed (Participants) | 12 | 12 | 13
  CD4+.PilA, Day 0 | 32.8 (43.6) | 60.5 (92.87) | 32.6 (48.69)
  CD4+.PilA, Day 60: number analyzed (Participants) | 16 | 11 | 15
  CD4+.PilA, Day 60 | 169.1 (150.22) | 110.2 (67.81) | 57.1 (99.26)
  CD4+.PilA, Day 90: number analyzed (Participants) | 16 | 11 | 13
  CD4+.PilA, Day 90 | 508.6 (474.31) | 330.5 (412.4) | 99 (152.45)
  CD4+.PilA, Day 210: number analyzed (Participants) | 7 | 9 | 11
  CD4+.PilA, Day 210 | 326 (208.31) | 220.8 (148.59) | 43.7 (69.03)
  CD4+.PilA, Day 420: number analyzed (Participants) | 10 | 8 | 12
  CD4+.PilA, Day 420 | 348.8 (376.87) | 131.1 (75.89) | 59.1 (53.4)
  CD4+.UspA2, Day 0: number analyzed (Participants) | 11 | 12 | 13
  CD4+.UspA2, Day 0 | 115.4 (154.96) | 126.3 (97.92) | 131.1 (182.97)
  CD4+.UspA2, Day 60 | 383.9 (326.2) | 253 (202.76) | 278.7 (672.84)
  CD4+.UspA2, Day 90: number analyzed (Participants) | 16 | 11 | 13
  CD4+.UspA2, Day 90 | 1392.6 (1145.48) | 979.2 (807.03) | 143.5 (237.29)
  CD4+.UspA2, Day 210: number analyzed (Participants) | 13 | 11 | 15
  CD4+.UspA2, Day 210 | 582.9 (376.54) | 322.8 (273.5) | 143.9 (242.72)
  CD4+.UspA2, Day 420: number analyzed (Participants) | 14 | 10 | 14
  CD4+.UspA2, Day 420 | 723.2 (763.51) | 385.4 (174.08) | 126.6 (187.52)

20. Secondary Outcome: Frequency of Specific CD8+ T-cells Against NTHi-Mcat Antigens Collected for the Evaluation of Cell-mediated Immune Response
Description: Frequency of specific CD8+ T-cells are measured by flow cytometry intracellular cytokine staining (ICS) expressing two or more markers (such as IL-2, IL-13, IL-17, IFN-γ, TNF-α and CD40L). The frequency of specific CD8+ T-cells are summarised [descriptive statistics: Mean and standard deviation (SD)] against each antigen (PD, PE, PilA and UspA2), by group in Step 2 at each time point during which blood samples are collected for CMI.
Time Frame: At Day 0 (pre-dose 1); at Day 60 (post-dose 1); at Day 90, Day 210 and Day 420 (post-dose2).
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: CD8+ T-cells/million cells
Arm/Group | GSK3277513A F2 Group | GSK3277513A F3 Group | PLACEBO Group
Number analyzed (Participants) | 15 | 12 | 13
CD8+ T-cells/million cells
  CD8+.PD, Day 0: number analyzed (Participants) | 11 | 12 | 13
  CD8+.PD, Day 0 | 66 (88.69) | 27.9 (80.68) | 46.9 (73.28)
  CD8+.PD, Day 60: number analyzed (Participants) | 15 | 11 | 12
  CD8+.PD, Day 60 | 29.4 (49.67) | 1 (0) | 20.5 (55.1)
  CD8+.PD, Day 90: number analyzed (Participants) | 14 | 10 | 12
  CD8+.PD, Day 90 | 66.5 (97.16) | 7.7 (21.19) | 49 (64.89)
  CD8+.PD, Day 210: number analyzed (Participants) | 11 | 12 | 11
  CD8+.PD, Day 210 | 66.4 (101.79) | 16.8 (42.84) | 17.7 (33.01)
  CD8+.PD, Day 420: number analyzed (Participants) | 13 | 8 | 12
  CD8+.PD, Day 420 | 43.2 (51.32) | 10.6 (17.98) | 37.3 (70.58)
  CD8+.PE, Day 0: number analyzed (Participants) | 11 | 12 | 12
  CD8+.PE, Day 0 | 42.4 (52.5) | 33.3 (59.32) | 74.4 (175.42)
  CD8+.PE, Day 60: number analyzed (Participants) | 15 | 11 | 12
  CD8+.PE, Day 60 | 27.8 (46.77) | 26.1 (40.81) | 42.7 (107.03)
  CD8+.PE, Day 90: number analyzed (Participants) | 14 | 10 | 12
  CD8+.PE, Day 90 | 30.4 (52.48) | 19.8 (43.69) | 45.4 (82.76)
  CD8+.PE, Day 210: number analyzed (Participants) | 12 | 12 | 12
  CD8+.PE, Day 210 | 31.8 (52.08) | 30.6 (62.25) | 44.2 (85.37)
  CD8+.PE, Day 420: number analyzed (Participants) | 15 | 10 | 12
  CD8+.PE, Day 420 | 5.7 (10.89) | 27 (58.46) | 19.4 (44.74)
  CD8+.PilA, Day 0: number analyzed (Participants) | 11 | 12 | 13
  CD8+.PilA, Day 0 | 34.6 (57.02) | 16 (40.27) | 44.7 (58.58)
  CD8+.PilA, Day 60: number analyzed (Participants) | 15 | 11 | 12
  CD8+.PilA, Day 60 | 26 (82.07) | 35.1 (39.81) | 28.7 (72.65)
  CD8+.PilA, Day 90: number analyzed (Participants) | 14 | 10 | 11
  CD8+.PilA, Day 90 | 50.8 (82.01) | 27.9 (43.03) | 28.3 (45.69)
  CD8+.PilA, Day 210: number analyzed (Participants) | 8 | 9 | 9
  CD8+.PilA, Day 210 | 11.3 (19.17) | 30.9 (70.04) | 21.4 (35.86)
  CD8+.PilA, Day 420: number analyzed (Participants) | 10 | 7 | 10
  CD8+.PilA, Day 420 | 28 (50.45) | 23 (37.7) | 28 (39.21)
  CD8+.UspA2, Day 0: number analyzed (Participants) | 10 | 12 | 13
  CD8+.UspA2, Day 0 | 22.5 (35.07) | 34.9 (50.24) | 85.3 (140.42)
  CD8+.UspA2, Day 60: number analyzed (Participants) | 15 | 11 | 12
  CD8+.UspA2, Day 60 | 29.3 (67.7) | 27.7 (50.12) | 21 (36.81)
  CD8+.UspA2, Day 90: number analyzed (Participants) | 14 | 10 | 11
  CD8+.UspA2, Day 90 | 74.1 (99.92) | 20.6 (26.17) | 37.4 (76.73)
  CD8+.UspA2, Day 210: number analyzed (Participants) | 13 | 11 | 13
  CD8+.UspA2, Day 210 | 61.5 (89.07) | 17.3 (26.54) | 48.1 (53.97)
  CD8+.UspA2, Day 420: number analyzed (Participants) | 15 | 10 | 12
  CD8+.UspA2, Day 420 | 16.7 (24.45) | 25.3 (70.42) | 48.8 (86.71)

ADVERSE EVENTS:
Time Frame: Solicited symptoms:within the 7-day post-vaccination period and Unsolicited AEs: during 30 days post- vaccination period. SAEs: during the whole study period (from Day 0 to Day 420)
Arm/Group | GSK3277513A F1 Group | GSK3277513A F2 Group | GSK3277513A F3 Group | PLACEBO Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/31 | 0/30 | 0/44
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/31 | 1/30 | 2/44
Other Adverse Events (participants affected / at risk) | 11/15 | 28/31 | 29/30 | 32/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3277513A F1 Group (N=15) | GSK3277513A F2 Group (N=31) | GSK3277513A F3 Group (N=30) | PLACEBO Group (N=44)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3277513A F1 Group (N=15) | GSK3277513A F2 Group (N=31) | GSK3277513A F3 Group (N=30) | PLACEBO Group (N=44)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 4 (6) | 10 (12) | 18 (24) | 12 (16)
Gastrointestinal disorder (Gastrointestinal disorders) | 4 (4) | 2 (2) | 5 (7) | 3 (4)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 7 (10) | 7 (8) | 16 (21) | 10 (13)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Injection site erythema (General disorders) | 0 (0) | 5 (6) | 5 (6) | 0 (0)
Injection site pain (General disorders) | 7 (9) | 25 (43) | 28 (51) | 11 (14)
Injection site swelling (General disorders) | 0 (0) | 5 (6) | 3 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymph gland infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 11 (15) | 12 (17) | 6 (7)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 5 (6) | 7 (10) | 11 (11)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (2) | 3 (3) | 5 (5) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Sterile pyuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-03-16): https://cdn.clinicaltrials.gov/large-docs/74/NCT02547974/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-06): https://cdn.clinicaltrials.gov/large-docs/74/NCT02547974/SAP_001.pdf